CLINICAL TRIAL: NCT05137886
Title: PD-1 Inhibitor Combined With Decitabine Followed by ASCT as Second-line Therapy for Relapsed or Refractory Classic Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Zou Dehui, Assistant Director of lymphoma Diagnosis and Treatment Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021051-EC-1
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Hodgkin Lymphoma, Adult; Relapse; Refractory Hodgkin Lymphoma
Keywords: Hodgkin lymphoma; relapse; refractory; autologous stem cell transplantation; PD-1 inhibitor; decitabine
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Immune Checkpoint Inhibitors; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 inhibitor combined with decitabine followed by ASCT (Experimental): Patients will receive salvage treatment of PD-1 inhibitor Tislelizumab combined with decitabine for four cycles, If PR or CR was obtained after salvage treatment, patients will receive GBM (gemcitabine, bulsufan and melphalan) conditioning regimen followed by ASCT. High-risk patients will receive PD-1 inhibitor for 1 year after ASCT as maintenance therapy.
  Interventions: Drug: PD-1 inhibitor

INTERVENTIONS:
Drug: PD-1 inhibitor — decitabine 10mg on d1-5, Tislelizumab 200mg on d8，21 days as one cycle.
  Other Names: decitabine; autologous stem cell transplantation

SUMMARY:
Young patients with relapsed or refractory classic Hodgkin's lymphoma will be treated with PD-1 inhibitor combined with decitabine as second-line salvage treatment for four cycles. If PR or CR was obtained after salvage treatment, patients will receive GBM conditioning regimen followed by ASCT as consolidation therapy. High-risk R/R cHL patients will be treated with PD-1 inhibitor after ASCT for 1 year. The purpose of current study is to determine the clinical efficacy and safety of PD-1 inhibitor combined with decitabine followed by ASCT as second-line treatment in patients with relapsed or refractory classic Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histological confirmation of relapsed or refractory classic Hodgkin lymphoma (HL).
2. 18 to 65 years of age.
3. Subjects with lymphoma must have at least one measureable lesion >1 cm as defined by lymphoma response criteria.
4. Proper functioning of the major organs: 1) The absolute value of neutrophils (≥1×10^9/L); 2) platelet count (≥75×10^9/L); 3) Serum creatinine <1.5 times Upper Limit Normal (ULN) ; 4) Serum total bilirubin < 1.5 times ULN; 5) Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) ≤3 times ULN; 6) Serum creatinine (Cr) ≤2 ULN, or glomerular filtration rate ≥40ml/min; 7) Thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were all within the normal range (±10%).
5. Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
6. LVEF value measured by echocardiography ≥50%.
7. Life expectancy > 3 months.

Exclusion Criteria:

1. Patients with central nervous system involvement by lymphoma.
2. Patients with active autoimmune diseases requiring systematic treatment in the past two years (hormone replacement therapy is not considered systematic treatment, such as type I diabetes mellitus, hypothyroidism requiring only thyroxine replacement therapy, adrenocortical dysfunction or pituitary dysfunction requiring only physiological doses of glucocorticoid replacement therapy); Patients with autoimmune diseases who do not require systematic treatment within two years can be enrolled.
3. Known systemic vasculitides, primary or secondary immunodeficiency(such as HIV infection or severe inflammatory disease).
4. Pregnant or breastfeeding women.
5. Major surgery within 4 weeks before enrollment.
6. Impaired cardiac function:Ejection fraction <50% on MUGA scan. QTc interval > 450msecs on baseline ECG. Myocardial infarction within 6 months prior to starting study; other clinically significant heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension, uncontrolled arrhythmias).
7. Other concurrent severe and/or uncontrolled medical conditions: Patients with another primary malignant disease, except those that do not currently require treatment; acute or chronic liver, pancreatic or severe renal disease; another severe and/or life-threatening medical disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  PFS

SECONDARY OUTCOMES:
Objective response rate | 2 years
  ORR
Complete response rate | 2 years
  CRR
Duration of response | 2 years
  DOR
Overall survival rate | 2 years
  OS
Severity of the adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided